CLINICAL TRIAL: NCT04182906
Title: Pediatric ACEs Screening and Resiliency Study
Acronym: PEARLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2016-089
Record Dates: First submitted 2019-11-19; First posted 2019-12-02 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Fibrinogen Abnormality; Telomere Length, Mean Leukocyte; Atopic; Acute Infection; Inflammatory Response; Self-regulation
Keywords: Adverse Childhood Experiences; Trauma; Social Determinants of Health; Child Mental Health; Resiliency; Primary Care; Universal screening
MeSH Terms: conditions — Self-Control; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be randomized twice. The first randomization will result in 3 arms (No ACEs screen, Identified ACEs screen, De-Identified ACEs screen). Participants in the No ACEs screen group or who screen ACEs=0 will receive care as usual. The second randomization will occur for those who screen with ACEs => 1, into two treatment groups (Care Coordination or Resiliency Clinic).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No ACEs screen (Active Comparator): Participants complete all measures except an ACEs screening tool
  Interventions: Behavioral: Usual Care
- Identified ACEs screen with Anticipatory Guidance (Experimental): Caregiver-completed screening tool about child's adverse experiences.In this version, specific ACEs items are reported, Pediatric medical provider offers anticipatory guidance about ACEs and toxic stress.
  Interventions: Behavioral: Care Coordination; Behavioral: Resiliency Clinic
- De-Identified ACEs screen with Anticipatory Guidance (Experimental): Caregiver-completed screening tool about child's adverse experiences. In this version,total number of ACEs items are reported, only. Pediatric medical provider offers anticipatory guidance about ACEs and toxic stress.
  Interventions: Behavioral: Care Coordination; Behavioral: Resiliency Clinic

INTERVENTIONS:
Behavioral: Care Coordination — Screening and referral for basic needs and adult mental health
  Arms: De-Identified ACEs screen with Anticipatory Guidance; Identified ACEs screen with Anticipatory Guidance
Behavioral: Resiliency Clinic — Mindfulness-based caregiver-child group medical care
  Arms: De-Identified ACEs screen with Anticipatory Guidance; Identified ACEs screen with Anticipatory Guidance
Behavioral: Usual Care — Usual Primary Pediatric Care
  Arms: No ACEs screen

SUMMARY:
Stressful and traumatic experiences in childhood (Adverse Childhood Events, or ACEs) have been associated with poor health outcomes that extend into adulthood. When stress is sustained or severe in the absence of an adequate buffer, the stress response can become dysregulated--a state referred to as toxic stress. Some professional organizations have advocated for ACEs screening to be part of routine medical care. To date, however, no ACEs screening tool has been validated for use with children. Intervening early at critical points in the life course has the potential to allow a child to avoid the negative consequences of these adverse events.

The proposed study has three overarching aims: (1) Examine the relationship between ACEs, stress biomarkers, and symptoms in children and caregivers over time; (2) Validate an ACEs screening in a pediatric health care setting; and (3) Test whether providing primary care-based preventive interventions for children with or at risk for toxic stress can lead to detectable changes in biomarkers, behavior, or health outcomes for children and/or caregivers.

DETAILED DESCRIPTION:
The study first aims to validate a pediatric ACEs screening tool. The creation of a scientifically validated, standard screening tool is a crucial step that will facilitate widespread screening for ACEs in clinical pediatric settings.

Subject participants will be randomized to either a control group or to an ACEs screening group. For the ACEs screening group, participants will be further randomized to 2 different formats for screening: (1) identified screening in which each individual item is endorsed or (2) de-identified screening in which only a total composite score is known.

Universal screening has limited utility in the absence of effective long-term interventions, and to date there are limited evidence-based interventions for the physiological and physical health consequences of toxic stress. This study will provide all families with ACEs-specific anticipatory guidance. Families with one or more ACEs will then be randomized to one of two interventions: Care Coordination or a Resiliency Clinic. Both of these interventions will specifically address ACEs-related needs, and will be evaluated based on mental and physical health outcomes as well as biomarker profiles before and after the intervention.

Care coordination will be based on the Family Information & Navigation Desk (FIND) Program model as implemented at UCSF Benioff Children's Hospital Oakland. The overarching goal of care-coordination is to routinely identify a family's basic social needs, in this case based on ACEs screener results, and then connect the family to appropriate community resources. This model moves beyond a focus on biomedical and risk-behavior explanations of health to understand the root causes of health inequities and provides a preventive approach to population health. The goal is to target the social and environmental factors that profoundly impact health.

The Resiliency Clinic will be an innovative monthly, mindfulness-based, caregiver-child group intervention focused on understanding toxic stress, and the development of self-regulation and co-regulation skills in caregivers and children identified as exposed to ACEs. The curriculum is based on existing models of mindfulness intervention and the structure of the caregiver-child group will be based upon 30 years of experience at UCSF Benioff Children's Hospital Oakland's Early Intervention Services, with group collaboration from pediatric medical providers, developmental and behavioral specialists, and mental health specialists.

The entire research project will be anchored by the collection of bio-specimens on each child. The normal stress response to acute life events induces several physiological responses that aid in adaptation and survival. Chronic exposure to adversity may result in a disruption of these normal stress pathways and is known as the toxic stress response (TSR). Several pathways have been suggested and include inflammatory and non-inflammatory mechanisms (disrupted neuroendocrine and/or autonomic nervous system functioning), epigenetic modification, and alteration of the body's microbiome. These pathways are sensitive to individual differences and adaptation mechanisms and aberrations in any of these pathways may negatively affect disease outcomes. An increased understanding of the multiple pathways of stress may unveil causal mechanisms that can lead to novel clinical interventions and allow for better targeting of these interventions. The biomarkers selected for this proposal are representative of the hypothesized pathways to disease and were selected based on relevance, clinical availability, and novelty. The collection of bio-specimens on all patients enrolled in the study will deepen our understanding of the correlations between ACEs, stress physiology and health outcomes. It will ground all aspects of this project in the underlying bio-chemical and genetic links between adversity and health outcomes. Biomarkers may help evaluate the concurrent validity of the pediatric ACEs screening tool and may offer insight on the pathways to poor health outcomes as a result of exposure to ACEs. Evaluating biomarker patterns and health outcomes in relation to ACE scores may allow for the establishment of a meaningful threshold for a clinical cut-point to the ACE score. Measuring biomarkers and therefore stress physiology before and after interventions may lead to more targeted and appropriate referrals and treatment modalities.

Ultimately, this study will help advance ACE screening in the pediatric clinic setting, offer families and providers further direction in choosing ACEs-related interventions, provide insight into the underlying biochemical patterns associated with adverse childhood experiences, and lay a strong foundation for future work elucidating the specific underlying mechanisms causing childhood adversity to lead to poor mental and physical health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* English and Spanish-speaking
* Patients receiving a well visit at Primary Care.
* Parents/primary caregivers of the children above, ages 18 and over, who are also legal guardians capable of consent.

Exclusion Criteria:

* Children who are dependents of the court
* Caregiver active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with full participation in the study
* Child or caregiver serious illness (mental or physical; requiring systemic treatment and/or hospitalization) or significant developmental disability that would interfere with full participation in the study
* Inability or unwillingness of subject or legal guardian/representative to give written informed consent.

Ages: 3 Months to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 555 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Validate a social determinants of health and adverse childhood experiences Screening tool | 12 months
  Determine the best format of screening either identified (each question individually is answered) vs de-identified (only a total composite score is known) for adverse childhood experiences using the PEARLS (Pediatric Early Adversity and Related Life Advent Screen) tool.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Global scale | 12 months
  Caregiver report of child global health with the PROMIS 10-item global health scale (t-scores 0-100; higher score = better global health)
Behavioral Rating Inventory of Executive Functioning (BRIEF 2/P) | 12 months
  Caregiver report of child executive functioning with the BRIEF-2/P questionnaire (t scores 0-100' higher scores are indicative of executive functioning issue, 65 or high is clinical threshold)
International Study of Asthma and Allergies in Childhood Questionnaire (ISSAC) | 12 months
  Validated instrument that assesses caregiver report of child asthma, allergic rhinitis and atopic dermatitis. Presence of the conditions is coded as yes/no variable.
Body mass index | 12 months
  Child body mass index calculated from measurement of height and weight (BMI = kg/m2 ). Higher BMI can be indicative of an issue above established threshold based on age and sex.

OTHER OUTCOMES:
Perceived Stress Scale (PSS) | 12 months
  Caregivers self-report on their perception of stress using the four-item Perceived Stress Scale (PSS). Range of scores 0-16; higher scores indicative of greater perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Dayna Long, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland; Neeta Thakur, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Benioff Children's Hospital Oakland, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Thakur N, Hessler D, Koita K, Ye M, Benson M, Gilgoff R, Bucci M, Long D, Burke Harris N. Pediatrics adverse childhood experiences and related life events screener (PEARLS) and health in a safety-net practice. Child Abuse Negl. 2020 Oct;108:104685. doi: 10.1016/j.chiabu.2020.104685. Epub 2020 Sep 5. PMID 32898839
- [Derived] Long D, Hessler D, Koita K, Bucci M, Benson M, Gilgoff R, Thakur N, Burke Harris N. Screening for adverse childhood experiences in pediatrics: A randomized trial of aggregate-level versus item-level response screening formats. PLoS One. 2022 Dec 15;17(12):e0273491. doi: 10.1371/journal.pone.0273491. eCollection 2022. PMID 36520927